CLINICAL TRIAL: NCT05285917
Title: BrUOG 419 - Promoting Utilization and Safety of Hydroxyurea Using Precision in Africa (PUSHUP)
Brief Title: Promoting Utilization and Safety of Hydroxyurea Using Precision in Africa
Acronym: PUSHUP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 419; U01HL157872 (NIH)
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Anemia in Children; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Weight Based Starting Dose (Active Comparator): 25 mg/kg starting dose Hydroxyurea
  Interventions: Drug: Hydroxyurea
- PK-guided starting dose (Experimental): Individualized, PK-guided starting dose Hydroxyurea
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea has a narrow therapeutic window such that selection of the correct dose is essential to optimize benefits and avoid toxicity.
  Other Names: Hydrea; Droxia

SUMMARY:
Sickle cell anemia (SCA) is among the world's most common and devastating blood disorders, affecting more than 300,000 newborns per year. Most infants with SCA are born in the low-resource settings of sub- Saharan Africa, where an estimated 50-90% will die before 5 years of age due to lack of early diagnosis and appropriate care. Hydroxyurea is a safe and effective once-daily oral medication that has become the standard of care for the treatment of children with SCA in high-resource settings. There is now a growing body of evidence to support the safety and clinical benefits of hydroxyurea for the treatment of SCA in sub-Saharan Africa. The requirement for frequent laboratory monitoring, uncertainties about appropriate, most effective dosing, and the concern for hematologic laboratory toxicities, however, will continue to limit widespread hydroxyurea utilization and real-world effectiveness. The investigators have recently developed and prospectively evaluated an individualized, pharmacokinetics-guided hydroxyurea dosing strategy for children with SCA that has demonstrated optimal clinical and laboratory benefits with minimal toxicity. In this research study, the investigators aim to extend this precision medicine approach to Africa.

DETAILED DESCRIPTION:
The Promoting Utilization and Safety of Hydroxyurea Using Precision in Africa (PUSHUP) trial is a prospective, randomized clinical trial of hydroxyurea for 400 children with SCA in Luanda, Angola. The study will prospectively evaluate the safety and efficacy of hydroxyurea with limited laboratory monitoring and will bring precision medicine to children with SCA using several novel features including measurement of hydroxyurea using a battery-powered HPLC machine and individualized dose calculations using an automated computer-based algorithm. The objective of this study is to establish evidence-based guidelines for hydroxyurea in sub-Saharan Africa, including appropriate dosing and laboratory monitoring strategy with the goal of allowing for widespread use of hydroxyurea across sub-Saharan Africa, regardless of clinical or laboratory resources.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell anemia (HbSS or HbS/B0-thalassemia)
* Age 6 months- 12 years of age at enrollment
* Parent or guardian willing and able to provide written or informed consent
* Weight ≥ 7.5 kg (temporary exclusion)

Exclusion Criteria:

* Splenomegaly with evidence of hypersplenism as defined by platelet count <150,000, hemoglobin <5 g/dL or absolute neutrophil count <1.0 x10^9/L
* Hydroxyurea use within the past 6 months
* Blood transfusion within the past 6 months (temporary exclusion)
* Pregnancy
* Pre-existing severe hematologic toxicity, as defined by platelet count <80,000, hemoglobin <4 regardless of ANC; hemoglobin <6 AND ARC <100; hemoglobin <7 AND ARC <80 x10^9/L (temporary exclusion)

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical, sickle cell adverse events (grade ≥ 3) as assessed by CTCAE v5.0 | From start of study treatment through first 12 months of treatment.
  These events will primarily include vaso-occlusive painful events, acute chest syndrome, stroke, acute splenic sequestration, and death. Data regarding adverse events, including severity grade and relatedness to SCA will be determined on site by the local investigator. All events will be centrally adjudicated by a blinded hematologist who is not a primary study investigator (Medical Safety Monitor) for inclusion in this endpoint.
Number of non-SCA related adverse events (grade ≥3), including death as assessed by CTCAE v5.0 | From start of study treatment through treatment completion, approximately 24 months.
  The clinical event rate with limited laboratory monitoring will be compared to the 3-months prior to hydroxyurea therapy.

SECONDARY OUTCOMES:
Hematologic response at 12 months | From start of study treatment through first 12 months of treatment.
  As measured by %HbF, proportion of participants in each arm with HbF ≥ 30%, hemoglobin, absolute reticulocyte count, absolute neutrophil count, platelet count, and mean corpuscular volume), hematologic laboratory toxicities (dose limiting toxicities defined a priori), hospitalizations, death, and all adverse events grade ≥ 3 (SCA and non-SCA related) as assessed by CTCAE v5.0.

OTHER OUTCOMES:
Health-Related Quality of Life Questionnaires | From start of study treatment through treatment completion, approximately 24 months.
  To evaluate the utility and validity of two established measures of health-related quality of life (HRQoL) for patients and families affected by SCA in Angola before and after hydroxyurea treatment. we will evaluate the Pediatric Quality of Life Sickle Cell Disease (PedsQL SCD) module for children ≥ 2 years of age and the PedsQL™ Family Impact Module for families of all enrolled participants. We will also utilize the International Sickle Cell World Assessment Survey (SWAY). These tools are available in the Portuguese language; for consistency and to account for the likely low literacy rate in the population, all surveys will be administered verbally to participants by study staff, recorded on paper or via tablet. We will compare results before and after hydroxyurea treatment. We will compare results to each other and to the published literature from other SCA populations.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T McGann, MD, MS, Principal Investigator — Rhode Island Hospital and Hasbro Children's Hospital
Locations (1):
- Hospital Geral dos Cajueiros, Luanda, Angola

IPD SHARING:
Plan to Share IPD: No